CLINICAL TRIAL: NCT05107622
Title: Administration of L. Paracasei 28.4 as an Adjunct to the Treatment of Periodontitis: Superiority Placebo-controlled Randomized Clinical Trial
Brief Title: Administration of L. Paracasei 28.4 as an Adjunct to the Treatment of Periodontitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Associate Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lp + PD
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMUD+Probiotic (Experimental): FMUD+Probiotic (n=30): full-mouth ultrasonic periodontal debridement associated with administration of probiotic formulation twice a day for 30 days.
  Interventions: Other: FMUD+Probiotic
- FMUD+Placebo (Placebo Comparator): FMUD+Placebo (n=30): full-mouth ultrasonic periodontal debridement associated with administration of placebo formulation, twice a day for 30 days.
  Interventions: Other: FMUD+Placebo

INTERVENTIONS:
Other: FMUD+Probiotic — Full-mouth ultrasonic periodontal debridement associated with administration of probiotic formulation (Lactobacillus paracasei 28.4) twice a day for 30 days.
  Arms: FMUD+Probiotic
Other: FMUD+Placebo — Full-mouth ultrasonic periodontal debridement associated with administration of placebo formulation twice a day for 30 days.
  Arms: FMUD+Placebo

SUMMARY:
The aim of this study is to evaluate the effects of probiotic administration of L. paracasei 28.4 as an adjunct to the non-surgical periodontal treatment in patients with periodontitis.

DETAILED DESCRIPTION:
This is a superiority placebo-controlled randomized clinical trial. The population that will be evaluated in the study will be selected at Institute of Science and Technology (ICT), São José dos Campos, College of Dentistry.

Sixty patients presenting Stage III/IV and Grade B/C periodontitis will be divided into 2 groups:

* FMUD+Placebo (n=30): full-mouth ultrasonic periodontal debridement associated with administration of placebo formulation, twice a day for 30 days;
* FMUD+Probiotic (n=30): full-mouth ultrasonic periodontal debridement associated with administration of probiotic formulation twice a day for 30 days.

The study will consist of two stages of treatment:

* Initial therapy: Before starting treatment, a complete examination of the oral cavity and evaluation of periodontal parameters will be performed. All patients will undergo a prior adjustment of the oral environment and oral hygiene. Thirty days after completion of initial therapy, a new periodontal evaluation will be performed and only patients who present a visible plaque index less than or equal to 25% will undergo subgingival periodontal debridement.
* Non-surgical periodontal therapy: After initial therapy, all patients will receive full-mouth ultrasonic periodontal debridement. Debridement will be performed by a single operator, trained, blind to the allocation of patients and different from the evaluator. If there is any complication that prevents the completion of full-mouth debridement, the procedure will be finished within a maximum period of 24 hours. The randomization envelope will be opened and the probiotic/placebo formulation will be delivered to patients. They will be instructed to consume the samples twice a day during the 30 days following periodontal treatment.

All clinical measurements will be performed by a single researcher, previously calibrated for the measurements. After periodontal therapy, treatment results will be evaluated three and six months after periodontal debridement associated with the use of placebo/probiotic formulation. Indications of adverse oral effects will be verified by visual assessment at 7, 30 and 90 days after the start of consumption of formulations.

To assess patient-centered parameters, the OHIP-14 questionnaire will be applied before and after 6 months of periodontal treatment for each patient. A 30-days diary will be used to assess the adherence to use and occurrence adverse effects.

Microbiological and immunological analyzes will be carried out through subgingival biofilm and gingival crevicular fluid samples collected from sites with moderate pockets and sites with deep pockets at baseline, 3 and 6 months after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III/IV and grade B/C generalized periodontitis;
* Presence of at least 20 teeth in the mouth;
* Signing the informed consent form.

Exclusion Criteria:

* Presence of systemic conditions that contraindicate the periodontal procedure or influence the progression of the disease;
* Periodontal treatment history in the last six months;
* Use of antibiotics or probiotics in the last six months;
* Smoke more than 10 cigarettes a day;
* Pregnant or breastfeeding;
* Chronic use of anti-inflammatory drugs or medications that can alter the response of periodontal tissues;
* Need of antibiotic prophylaxis for dental procedures;
* Need of probiotic therapy.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Number of pockets with PD ≥ 5 mm | 6 months
  Number of pockets with probing depth ≥ 5 mm

CONTACTS AND LOCATIONS:
Overall Officials: Laís F Ferraz, MS, Principal Investigator — Sao Paulo State University - Brazil; Mauro P Santamaria, PhD, Study Director — Sao Paulo State University - Brazil
Locations (1):
- Mauro Pedrine Santamaria, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the end of the study after a direct request.
Supporting Information: Study Protocol, ICF
Time Frame: After the study completion.

REFERENCES:
- [Background] Ribeiro FC, Junqueira JC, Dos Santos JD, de Barros PP, Rossoni RD, Shukla S, Fuchs BB, Shukla A, Mylonakis E. Development of Probiotic Formulations for Oral Candidiasis Prevention: Gellan Gum as a Carrier To Deliver Lactobacillus paracasei 28.4. Antimicrob Agents Chemother. 2020 May 21;64(6):e02323-19. doi: 10.1128/AAC.02323-19. Print 2020 May 21. PMID 32253208
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Background] Teughels W, Durukan A, Ozcelik O, Pauwels M, Quirynen M, Haytac MC. Clinical and microbiological effects of Lactobacillus reuteri probiotics in the treatment of chronic periodontitis: a randomized placebo-controlled study. J Clin Periodontol. 2013 Nov;40(11):1025-35. doi: 10.1111/jcpe.12155. Epub 2013 Sep 15. PMID 24164569